CLINICAL TRIAL: NCT03045549
Title: Home-based Rehabilitation With A Digital Biofeedback System Versus Conventional Rehabilitation After Total Hip Replacement: a Pilot Study
Brief Title: Digital Biofeedback System Versus Conventional Home-based Rehabilitation After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Collaborators: Hospital da Prelada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH-THR-01
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hip Osteoarthritis; Hip Arthrosis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All patients will be assessed for clinical outcomes by an independent rater blinded to the study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Home-based rehabilitation sessions performed with the digital biofeedback system. Patients will be instructed to perform exercise sessions at least 5 days a week, but compliance to this schedule is not mandatory.
  Interventions: Device: Digital biofeedback system
- Conventional rehabilitation group (Active Comparator): Home-based rehabilitation sessions provided by a Physical Therapist, 3 times a week, each with 1h duration. Patients will be instructed to perform 2 additional unsupervised sessions per week, but compliance to these sessions is not mandatory.
  Interventions: Other: Conventional home-based rehabilitation

INTERVENTIONS:
Device: Digital biofeedback system — The system will be used independently by the patients to perform rehabilitation sessions at home, under remote monitoring from the clinical team. A tailored rehabilitation program will be prescribed, based on the following principles:
  STAGE 1 (Weeks 0-6) Open kinetic chain exercises without added resistance: lying, sitting and standing (with support) Strengthening of hip flexors and abductors (mainly) Ice pack application STAGE 2 (weeks 7-8) Open kinetic chain exercises with added resistance: lying, sitting (high chair) and standing (with progression to standing without support) Strengthening of hip flexors and abductors (mainly) Ice pack application after each session
  Other Names: SWORD Phoenix
  Arms: Experimental group
Other: Conventional home-based rehabilitation — Patients will perform 3 weekly rehabilitation sessions, with a duration of 1 hour, for 8 weeks, provided by a physical therapist. The rehabilitation program will respect the following principles:
  STAGE 1 (Weeks 0-6) Soft tissue massage Active assisted mobilization of the hip joint to increase range of motion (avoiding internal rotation and adduction) Gait training with bilateral assistive devices Isometric exercises progressing to open chain, low-impact, concentric exercises with strengthening of hip abductors and flexors Ice pack application STAGE 2 (weeks 7-8) Soft tissue massage Gait training with progressive withdrawal of assistive devices Balance exercises with progression to one-leg support Open-chain strengthening exercises against resistance with progression to closed-chain exercises Ice pack application
  Arms: Conventional rehabilitation group

SUMMARY:
The study was designed to compare the clinical outcomes of a home-based rehabilitation program using a novel digital biofeedback system against conventional home-based rehabilitation after total hip replacement This system allows the patients to perform independent rehabilitation sessions at home, under remote monitoring from the clinical team. The investigators hypothesise that the clinical outcomes of a home-based rehabilitation program will be at least similar to the outcomes of a traditional home-based rehabilitation with face-to-face sessions. This is a single-center, prospective, parallel-group pilot study with active comparator. Patients will be enrolled pre-operatively and then divided into 2 groups: experimental group and conventional rehabilitation group. Both groups will perform an 8-week rehabilitation program starting between day 7 and 10 after surgery.

The experimental group will perform daily exercise sessions at home using the system, under remote monitoring from a physical therapist. The conventional rehabilitation group will perform 3 home-based rehabilitation sessions per week, each with 1h duration, given by a physical therapist.

Outcomes will be measured at weeks 4 and 8 and then at 3 and 6 months. The primary outcome is the change in patient performance measured by the Timed-up-and-Go (TUG) test between in comparison with the pre-operative score. Secondary outcomes will be measured in terms of: a) Hip Osteoarthritis Outcome Score (HOOS); b) range of motion of the hip joint (lying flexion/abduction; standing flexion/adbuction/hyperextension)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Clinical and imaging evidence of hip osteoarthritis
* Indication for total hip replacement according to the patient´s orthopedic surgeon
* Ability to walk unaided, with unilateral or bilateral support
* Availability of a carer to assist the patient after surgery

Exclusion Criteria:

* Patients admitted for revision of total hip replacement
* Contralateral hip or knee osteoarthritis severely limiting patient mobility and ability to comply with a rehabilitation program
* Aphasia, dementia or psychiatric comorbidity interfering with the communication or compliance to the rehabilitation process
* Respiratory, cardiac, metabolic or other condition incompatible with at least 30 minutes of light to moderate physical activity
* Major medical complications occurring after surgery that prevent the discharge of the patient within 7 days after the surgery
* Other medical and/or surgical complications that prevent the patient from complying with a rehabilitation program
* Blind and/or illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Change in the Timed Up and Go Test score | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  The timed up and go requires a patient to rise from a chair walk three meters around a piece of tape and return to the chair again as quickly as possible.

SECONDARY OUTCOMES:
Change in Hip injury and Osteoarthritis Outcome Score (KOOS) | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  The HOOS is a standardized and validated patient outcome score that assesses functional limitation in patients with hip problems.
Change in the Range of Motion (degrees) | Baseline; 4 and 8 weeks after initiation of rehabilitation program and then at 3 and 6 months after surgery
  Change in the hip range of motion (lying flexion/adbuction; standing flexion/abduction/hyperextension) measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — Sword Health, SA
Locations (1):
- Hospital da Prelada - Dr. Domingos Braga da Cruz, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon study publication, for 5 years.
Access Criteria: Study protocol will be available through a direct link in this platform. The excel file with the aggregate results will be made available as supplementary information upon study publication.

REFERENCES:
- [Derived] Dias Correia F, Nogueira A, Magalhaes I, Guimaraes J, Moreira M, Barradas I, Molinos M, Teixeira L, Pires J, Seabra R, Lains J, Bento V. Digital Versus Conventional Rehabilitation After Total Hip Arthroplasty: A Single-Center, Parallel-Group Pilot Study. JMIR Rehabil Assist Technol. 2019 Jun 21;6(1):e14523. doi: 10.2196/14523. PMID 31228176